CLINICAL TRIAL: NCT06949098
Title: An Exploratory Study of Local Resection Combined With Chemoradiotherapy in Patients With Low/Ultra-low Early-stage Rectal Cancer With a Strong Desire to Preserve the Anus
Brief Title: Tumor Local Excision +Postoperative Adjuvant Chemoradiotherapy for T1-2N0M0 Low/Ultra-Low Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025043
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer Stage I
Keywords: Adjuvant Chemoradiotherapy; Local excision; Low/ultra-low rectal cancer; Early rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Local Tumor Excision +Postoperative Adjuvant Chemoradiotherapy (Experimental): All enrolled patients will first undergo local tumor resection. Adjuvant therapy will be initiated 4-6 weeks postoperatively based on pathological staging:
  For pT1N0M0 patients without high-risk features:
  Active surveillance OR Radiotherapy alone (Prescription: Pelvic field irradiation 45Gy in 25 fractions)
  For pT2N0M0 or pT1N0M0 patients with adverse prognostic factors:
  Adjuvant chemoradiotherapy (Prescription:Pelvic field irradiation 45Gy in 25 fractions PLUS Local tumor bed boost 5.4Gy in 3 fractions；Concurrent chemotherapy: Oral capecitabine 825mg/m² twice daily)；For patients with positive margins after local excision: Re-excision followed by adjuvant chemoradiotherapy OR Dose-escalated chemoradiotherapy (Prescription: Pelvic field irradiation 45Gy in 25 fractions PLUS Local tumor bed boost 14.4Gy in 8 fractions)；
  For patients with staging > pT2N0M0:
  Total mesorectal excision (TME) Following treatment completion, patients will enter clinical follow-up surveillance.
  Interventions: Procedure: Local Tumor Resection; Radiation: Radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Procedure: Local Tumor Resection — All enrolled patients will first undergo local tumor resection.
Radiation: Radiotherapy — Pelvic field irradiation 45Gy in 25 fractions plus Local tumor bed boost 5.4Gy in 3 fractions.
  For patients with positive surgical margins after local resection, a radiotherapy boost (pelvic field 45Gy/25 fractions + tumor bed local boost 14.4Gy/8 fractions) can be given.
Drug: Chemotherapy — Concurrent oral capecitabine 825 mg/m² twice daily with radiotherapy

SUMMARY:
This study is a single-center, single-arm, prospective clinical trial designed to evaluate the efficacy of local excision followed by postoperative chemoradiotherapy in patients with early-stage low/ultra-low rectal cancer. The study plans to enroll 60 patients with T1-2N0M0 low/ultra-low rectal cancer.

DETAILED DESCRIPTION:
Baseline examnation: All enrolled patients in this study, in addition to routine laboratory and imaging examinations such as blood routine, blood biochemistry, serum tumor markers (Incl. CEA, CA-199, CA-724 β2-microglobulin, Ferroprotein), chest CT, abdominal and pelvic MRI, etc., were required to undergo KRAS, NRAS, BREF, PD-L1, MMR/MSS testings before surgery, and blood lymphocyte subgroups were analyzed before surgery.

All enrolled patients will first undergo local tumor resection. Adjuvant therapy will be initiated 4-6 weeks postoperatively based on pathological staging:

For pT1N0M0 patients without high-risk features:

Active surveillance OR Radiotherapy alone (Prescription: Pelvic field irradiation 45Gy in 25 fractions)

For pT2N0M0 or pT1N0M0 patients with adverse prognostic factors (including poorly differentiated histology, lymphovascular invasion, positive margins*, tumor infiltration beyond the outer third of the submucosal muscle layer（SM3 level）, or submucosal invasion >1mm):

Adjuvant chemoradiotherapy (Prescription:Pelvic field irradiation 45Gy in 25 fractions PLUS Local tumor bed boost 5.4Gy in 3 fractions；Concurrent chemotherapy: Oral capecitabine 825mg/m² twice daily)；For patients with positive margins after local excision: Re-excision followed by adjuvant chemoradiotherapy OR Dose-escalated chemoradiotherapy (Prescription: Pelvic field irradiation 45Gy in 25 fractions PLUS Local tumor bed boost 14.4Gy in 8 fractions)；

For patients with staging > pT2N0M0:

Total mesorectal excision (TME) Following treatment completion, patients will enter clinical follow-up surveillance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender
2. ECOG performance status 0-1
3. Biopsy-proven rectal adenocarcinoma
4. Distal margin of primary tumor ≤8 cm from anal verge
5. Clinical stage I (cT1-2N0M0)
6. Strong organ preservation preference with refusal to undergo abdominoperineal resection (Miles operation)
7. The surgeon determined a local resection was feasible
8. No contraindications to chemoradiotherapy

Exclusion Criteria:

1. Failure to meet the above inclusion criteria
2. Patients refusing to sign informed consent
3. Impaired cognitive function or psychiatric disorders
4. Patients deemed ineligible by investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
5-year DFS Rate | 5 years
  Defined as the proportion of subjects who remain free from recurrence, progression, or death for 5 years after completing surgery and adjuvant chemoradiotherapy (estimated as the proportion of event-free patients based on survival curves).

SECONDARY OUTCOMES:
5-year Local Recurrence Rate | 5 years
  The proportion of patients who experience tumor recurrence at or near the primary tumor site (within the pelvic region) within 5 years after initial treatment completion.
5-year Distant Metastasis Rate | 5 years
  The proportion of patients who develop metastatic disease in distant organs (e.g., liver, lungs, bones, or non-regional lymph nodes) within 5 years after initial treatment.
5-year OS | 5 years
  The proportion of patients who remain alive (regardless of disease status) at 5 years after initial diagnosis or treatment initiation.
Sphincter Retention Rate | 1 week after sugery
  The proportion of patients who successfully avoid permanent colostomy after rectal cancer treatment, maintaining natural anal sphincter function for defecation.
Quality of Life (QoL) Scores | 5 years
  Calculated based on standardized scores, with proportions of patients showing marked improvement, improvement, no change, or worsening. Specific calculation rules are provided in the appendix.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided